CLINICAL TRIAL: NCT06298812
Title: A Prospective, Single-Arm, Multi-Center, Registry Post-Approval Study of Growth Modulation in the Treatment of Idiopathic Scoliosis With the REFLECT™ Scoliosis Correction System
Brief Title: REFLECT Scoliosis System Post Approval Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Globus Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol Rev 0 11July2023
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Idiopathic Scoliosis

STUDY DESIGN:
Intervention Model Description: Patients treated with the REFLECT Scoliosis Correction System
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- REFLECT (Other): Enrolled patients are treated with the REFLECT Scoliosis System. This is an HDE-approved device.
  Interventions: Device: REFLECT Scoliosis Correction System

INTERVENTIONS:
Device: REFLECT Scoliosis Correction System — The REFLECT™ Scoliosis Correction System is designed for continued growth and mobility of the spine as well as straightening of the spine by holding the segments in a more natural anatomic position using non-rigid materials.

SUMMARY:
The purpose of this multi-center, prospective, single-arm registry Post-Approval Study (PAS) is to evaluate the radiographic and clinical outcomes of 100 patients with idiopathic scoliosis treated with the REFLECT™ Scoliosis Correction System, as a condition of HDE approval

DETAILED DESCRIPTION:
The REFLECT™ Scoliosis Correction System is designed for continued growth and mobility of the spine as well as straightening of the spine by holding the segments in a more natural anatomic position using non-rigid materials. REFLECT™ uses a growth modulation technique in which growth of the patient is used to achieve progressive scoliosis correction.

The REFLECT™ Scoliosis Correction System is indicated for skeletally immature patients who require surgical treatment to obtain and maintain correction of progressive idiopathic scoliosis, who have a major Cobb angle of 30 to 65 degrees whose osseous structure is dimensionally adequate to accommodate screw fixation, as determined by radiographic imaging. Patients should have failed bracing and/or are intolerant to brace wear.

A total of 100 patients will be prospectively enrolled and treated at a minimum of 5 U.S. sites, with a maximum of 20 subjects at any one site, with sequential enrollment from each site. Patients will be followed for 5 years with evaluations at the following timepoints: preoperative, intraoperative, immediate postoperative (first erect), 6 weeks, 6 months, 12 months, 24 months, and 60 months. Primary and secondary outcomes from 100 patients enrolled and treated with REFLECT™ will be summarized.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of progressive idiopathic scoliosis
* Preoperative major Cobb angle 30°-65°
* Preoperative flexibility to ≤30° on side bending radiograph (left or right)
* Skeletally immature at the time of surgery with Risser sign <5 or Sanders score <8
* Osseous structure dimensionally adequate to accommodate screw fixation, as determined by radiographic imaging
* Failed or intolerant to bracing
* Signed informed consent and/or assent forms specific to this study

Exclusion Criteria:

* Prior spinal surgery at the level(s) to be treated
* Documented poor bone quality, defined as a T-score of -1.5 or less
* Presence of any systemic infection, local infection, or skin compromise at the surgical site
* Any medical or surgical condition which would preclude the potential benefit of spinal surgery, such as coagulation disorders, allergies to the implant materials, and patient's unwillingness or inability to cooperate with post-operative care instructions
* Unwillingness, inability, or living situation (e.g. custody arrangements, homelessness, detention) that would preclude ability to return to the study site for follow-up visits as described in protocol and Informed Consent
* Active participation in a drug or device study that is more than minimal risk such that participation would confound the measurements of the present study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary Probable Benefit | 60 months postoperative
  Maintenance of major Cobb angle less than or equal to 40°
Primary Safety | 60 months postoperative
  Serious adverse events (SAEs) and device- or procedure-related adverse events (AEs)

SECONDARY OUTCOMES:
Curve progression | 60 months postoperative
  Curve progression no greater than 10° of any secondary curve above or below the implant, or development of a new curve equal to or greater than 40°
Device integrity | 60 months postoperative
  Device integrity failures including cord breakage and screw migration
Composite endpoint analysis | 60 months postoperative
  Maintenance of major Cobb angle less than or equal to 40° AND freedom from Serious Adverse Events (SAEs) during the procedure and procedure/device related SAEs following surgery
Failure analysis | 60 months postoperative
  Analysis of the failure attributable to conversion to another spinal implant OR major Cobb angle that exceeded 40° at defined follow-up visit OR any progression of the major curve at defined follow-up compared to baseline OR death OR permanent disability
SRS score | 60 months postoperative
  Mean score of Scoliosis Research Society 22r Patient Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No